CLINICAL TRIAL: NCT06746675
Title: Evaluating Healthy Families PrEP: an Intervention to Promote PrEP Use During Periconception, Pregnancy and Postpartum Periods for Women in Rural Uganda
Brief Title: Evaluating the Healthy Families PrEP Program for Women at Risk for HIV
Acronym: HFPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Lynn T. Matthews, Professor of Medicine Medicine, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300013932; R01MH134680 (NIH)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: HIV; Pregnancy; Pre-Exposure Prophylaxis of HIV Infection
Keywords: HIV; pregnancy; Pre-exposure prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Families PrEP Counselling Intervention (Active Comparator): Intervention Health Care Centers will offer the guideline-based PrEP standard of care plus trained staff will conduct the 3-session Healthy Families-PrEP intervention with HIV-uninfected women with plans for pregnancy in the next year and concerns about or exposure to HIV.
  Interventions: Drug: Healthy Families PrEP Counselling Intervention
- Standard of care PrEP services for perinatal women (No Intervention)

INTERVENTIONS:
Drug: Healthy Families PrEP Counselling Intervention — Healthy Families-PrEP intervention with HIV-uninfected women with plans for pregnancy in the next year and concerns about or exposure to HIV. Session 1 focuses on providing information about HIV prevention in the context of reproductive goals (using tools with locally developed images), increasing motivation for behavior change, and developing a safer conception plan (e.g., PrEP uptake, PrEP adherence, couples-based counselling and testing, delaying condomless sex until partner serostatus known and, if living with HIV, virally suppressed). Sessions 2 and 3 (conducted at 1 and 3 months) review the safer conception plan and revise as needed (e.g., changes in readiness to initiate PrEP, partner serostatus knowledge) and engaging in problem-solving barriers (including structural) to plan execution, communication skills training, and motivational strategies for successful plan execution. Participants receive quarterly adherence counseling using tools developed by this team.
  Arms: Healthy Families PrEP Counselling Intervention

SUMMARY:
Study investigators developed and piloted a counselling intervention, Healthy Families-PrEP, that supports women to use HIV prevention strategies while trying for and during pregnancy. They will now adapt the intervention to community clinics and postpartum women and test the intervention. The goal is to reduce HIV incidence among women and children.

DETAILED DESCRIPTION:
Women in Uganda who are planning for pregnancy, pregnant, or postpartum and have a partner living with HIV are vulnerable to acquiring HIV.

Adapting this intervention to community clinics and testing effectiveness aligns with global and Ugandan Ministry of Health goals to reduce HIV incidence among women of reproductive age and eliminate perinatal transmission. Additionally, costing analyses will be conducted to determine the cost of implementing HF-PrEP from both payer and societal perspectives. This work will inform future intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤45 years
* Willing and able to participate in the informed consent process
* HIV-uninfected by self-report, but have indications for HIV prevention strategies, such as having a partner living with HIV or who they think may be living with HIV
* Reporting pregnancy in the past 2 years, and/or desire to have a child in the next year, and/or have a partner who desires to a child in the next year
* Fluent in English or local language
* Living within 60km of a healthcare center included in the trial
* HIV Negative (onsite rapid testing)

Exclusion Criteria:

* Not reporting pregnancy in the past 2 years
* Does not report personal or partner desire to have a child in the next year
* Not willing to provide informed consent
* Not able to communicate in English or local language
* Does not report pregnancy in the past 2 years and/or does not report personal or partner desire to have a child in the next year
* Not able to communicate in English or local language
* Living beyond 60km of the trial healthcare center
* HIV-positive (onsite rapid testing)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with pregnancy intentions
Enrollment: 660 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation - Women who start to use PrEP | Enrolment to 6 months
  The primary effectiveness outcome will be proportion of women at 6 months with intracellular TFV-DP concentration consistent with taking at least 4 doses per week.

SECONDARY OUTCOMES:
Women who continue to use PrEP when they become pregnant | Enrolment to 18 months
  Investigators will explore secondary outcomes of PrEP adherence patterns over perinatal periods with quarterly blood draws for TFV measurements

CONTACTS AND LOCATIONS:
Overall Officials: Lynn T Matthews, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided